CLINICAL TRIAL: NCT07256613
Title: Outcomes of Non-surgical Periodontal Therapy on Urea and Creatinine Levels in Type-2 Diabetes Mellitus Patients
Brief Title: Non-surgical Periodontal Therapy and Kidney Outcomes in Type 2 Diabetes Mellitus
Acronym: KIDPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Ather Khan, Doctor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3642/DUHS/Approval/2024/311
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus MeSH:D003924; Periodontitis MeSH:D010518; Diabetic Nephropathies MeSH:D003928
Keywords: Type 2 Diabetes Mellitus; Uncontrolled Type 2 Diabetes; Diabetes-related nephropathy; Chronic kidney disease (CKD); Diabetic nephropathy; periodontitis; non surgical periodontal therapy; scaling; root palnning; serum creatinine; blood urea nitrogen; BUN; eGFR; MDRD GFR euation; oral hygiene instruction(OHI); Randomised control trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Diabetic Nephropathies; Periodontitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment - Participants are randomly assigned to one of two groups: an intervention group receiving non-surgical periodontal therapy and a control group receiving delayed therapy after the study period.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Surgical Periodontal Therapy (Scaling and Root Planing + Oral Hygiene Instructions) (Experimental): Participants in this arm will receive full-mouth non-surgical periodontal therapy, including ultrasonic scaling and manual root planing in a single session performed by trained dental hygienists. This treatment aims to remove supra- and subgingival plaque and calculus to reduce periodontal inflammation. Standardized oral hygiene instructions will also be provided, including demonstration of the Modified Stillman's brushing technique using a soft toothbrush and fluoridated toothpaste twice daily. Participants will be monitored for 90 days to assess changes in renal biomarkers (serum creatinine, blood urea nitrogen, and eGFR)
  Interventions: Procedure: scaling and root planning
- Control - Oral Hygiene Instructions with Delayed Periodontal Therapy (Active Comparator): Participants in the control arm will receive only standardized oral hygiene instructions at baseline and will not undergo scaling and root planing during the 90-day study period. After completion of follow-up assessments, they will receive the same periodontal therapy as the intervention group (delayed therapy) to ensure ethical equivalence
  Interventions: Procedure: scaling and root planning

INTERVENTIONS:
Procedure: scaling and root planning — Intervention 1: Scaling and Root Planing (SRP) + Oral Hygiene Instructions (OHI)
  Intervention Description:
  Participants assigned to the intervention arm will receive full-mouth non-surgical periodontal therapy consisting of scaling and root planning (SRP). Ultrasonic scalers will be used to remove supragingival plaque and calculus, followed by hand instruments (curettes and scalers) for subgingival debridement and root planing. The procedure is performed in a single session by trained and calibrated dental hygienists. Participants will also receive standardized oral hygiene instructions (OHI), including demonstration of the Modified Stillman's toothbrushing technique using a soft-bristle toothbrush and fluoridated toothpaste twice daily. Each participant will be provided with an oral hygiene kit to ensure consistency. Postoperative care includes warm saline rinses for three days. No further periodontal treatment will be given during the 90-day follow-up period.

SUMMARY:
Brief Summary (Lay Description)

This research study is being conducted to understand whether treating gum disease (periodontitis) can help improve kidney health in patients who have type-2 diabetes mellitus (T2DM). Both diabetes and gum disease are common long-term conditions that often occur together. People with uncontrolled diabetes are at risk of developing kidney problems due to damage in the small blood vessels of the kidneys - a condition known as diabetic nephropathy.

Scientific evidence has already shown that treating gum disease can help improve blood sugar control in diabetic patients. However, it is still unclear whether gum treatment can also help reduce the risk or severity of kidney-related complications. This study aims to find out if non-surgical periodontal therapy (NSPT), which includes scaling and root planing (deep dental cleaning), has any effect on blood markers of kidney function - specifically urea, creatinine, and estimated glomerular filtration rate (eGFR) - in patients with uncontrolled type-2 diabetes.

The study will be conducted as a randomized controlled trial involving 46 patients with uncontrolled T2DM (HbA1c ≥ 7%) who also have moderate to severe gum disease. Participants will be divided randomly into two groups:

Test Group: Will receive full-mouth non-surgical periodontal therapy (scaling and root planing) and oral hygiene instructions.

Control Group: Will receive oral hygiene instructions only and will get the same gum treatment later (after 90 days, as delayed therapy).

All participants will have their gum health examined, and blood tests will be done at the start and again after 90 days to measure urea, creatinine, and eGFR levels. These tests help determine how well the kidneys are working. The changes in these values before and after gum treatment will show whether improving oral health has any beneficial impact on kidney function in diabetics.

The study is expected to take one year and will be conducted at Dow University of Health Sciences, Karachi. All participants will receive standard dental and laboratory assessments at no cost. The results may help improve future strategies for managing diabetic patients by integrating oral health care with medical care.

Purpose:

To determine whether treating gum disease (through non-surgical periodontal therapy) can improve kidney function markers - urea, creatinine, and eGFR - in patients with uncontrolled type-2 diabetes mellitus.

Question being answered:

Does non-surgical periodontal therapy have a positive effect on kidney function in uncontrolled type-2 diabetic patients by reducing urea and creatinine levels and improving eGFR?

DETAILED DESCRIPTION:
Detailed Description Background and Rationale

Periodontitis and type 2 diabetes mellitus (T2DM) are both chronic, non-communicable diseases with a well-established bidirectional relationship. Individuals with poorly controlled diabetes are at higher risk of developing periodontal inflammation, while untreated periodontitis may contribute to poor glycemic control through systemic inflammation. Among the microvascular complications of diabetes, nephropathy remains a major cause of morbidity and mortality. It is characterized by glomerular damage, resulting in elevated serum creatinine (SCr) and urea levels, and a reduced glomerular filtration rate (GFR).

Although several studies have shown that periodontal therapy can improve glycemic control, there is limited evidence regarding its effects on renal function in diabetic patients. The systemic inflammatory burden caused by chronic periodontitis may exacerbate kidney dysfunction, as inflammatory mediators such as TNF-α, IL-1β, and prostaglandin E2 circulate systemically and contribute to endothelial damage. This study aims to evaluate whether non-surgical periodontal therapy (NSPT), by reducing periodontal inflammation and bacterial load, can positively influence renal biomarkers in patients with uncontrolled type 2 diabetes mellitus.

The study will provide preliminary interventional data on the potential of periodontal therapy as an adjunctive measure in reducing systemic inflammatory load and possibly delaying microvascular complications, such as diabetic nephropathy. This is particularly relevant in the Pakistani population, where both T2DM and periodontitis have high prevalence, yet local interventional evidence remains scarce.

Study Design and Setting

This is a parallel-arm, single-blinded randomized controlled clinical trial designed to evaluate the effect of NSPT on renal function markers in uncontrolled T2DM patients with moderate to severe periodontitis. The study will be conducted at two sites under Dow University of Health Sciences (DUHS), Karachi:

National Institute of Diabetes and Endocrinology (NIDE) - patient screening and medical evaluation.

Dr. Ishrat-ul-Ebad Khan Institute of Oral Health Sciences (DIKIOHS) - periodontal examination and intervention.

The total duration of the study is projected to be 12 months, including patient recruitment, intervention, 3-month follow-up, data analysis, and report preparation.

Sample Size and Allocation

Based on previous studies assessing serum creatinine differences between periodontitis and non-periodontitis groups, a sample size of 23 participants per arm (n=46 total) has been calculated, accounting for 20% attrition. Participants will be randomly assigned to one of two groups using computer-generated random numbers and allocation concealment via Serially Numbered Opaque Sealed Envelopes (SNOSE).

Test Group: Non-surgical periodontal therapy (scaling and root planing) + standardized oral hygiene instructions (OHI).

Control Group: OHI only; scaling and root planing provided after study completion as delayed therapy (DT).

The principal investigator will remain blinded to the intervention assignment during data collection and analysis.

Intervention Details

1. Non-Surgical Periodontal Therapy (NSPT)

   The NSPT intervention includes full-mouth ultrasonic scaling followed by manual root planing using Gracey curettes. This will be performed in a single session by trained and calibrated dental hygienists under supervision. The procedure aims to remove supra- and sub-gingival plaque and calculus, thereby eliminating bacterial niches contributing to inflammation.
2. Oral Hygiene Instructions (OHI)

   All participants will receive standardized instructions based on the Modified Stillman's brushing technique using a soft-bristle toothbrush and fluoridated toothpaste twice daily. Each participant will receive an identical oral hygiene kit to ensure standardization. Compliance will be monitored through self-maintained daily practice sheets reviewed at follow-up visits.
3. Delayed Therapy (DT)

Participants in the control arm will receive the same NSPT procedure after completion of the 90-day follow-up period to ensure ethical equivalence.

Clinical and Laboratory Assessments Baseline Examination

At recruitment, each participant will undergo:

Full-mouth periodontal charting (six sites per tooth) for probing depth (PPD), clinical attachment loss (CAL), and bleeding on probing (BOP).

Collection of demographic, medical, and lifestyle data via structured questionnaire.

Blood sampling for baseline measurement of:

Serum creatinine (SCr)

Blood urea nitrogen (BUN)

Glycated hemoglobin (HbA1c)

Estimated glomerular filtration rate (eGFR), calculated using the Modification of Diet in Renal Disease (MDRD) formula.

Follow-Up Examination

At 90 days post-intervention, all parameters will be re-evaluated to assess intra- and inter-group changes in renal and periodontal health indices.

Blood samples will be collected under aseptic conditions by trained personnel and analyzed by the Dow Diagnostic Laboratory using standardized procedures. Serum separation will be done by centrifugation; assays will follow clinical laboratory reference ranges:

SCr normal range: 0.6-1.5 mg/dL

BUN normal range: 30-40 mg/dL

Normal eGFR cutoff: ≥60 mL/min/1.73 m²

Calibration and Quality Control

All periodontal examinations will be performed by the principal investigator (PI), trained and calibrated against a gold standard examiner (the supervisor). Inter- and intra-examiner reliability will be tested before trial initiation using kappa statistics and intra-class correlation coefficients. The two dental hygienists performing the interventions will undergo calibration sessions to standardize SRP procedures. Random 10% re-evaluation of data will be done to ensure consistency.

Data Management and Statistical Analysis

All data will be anonymized using unique participant identifiers. Data entry will be performed using IBM SPSS version 26.0.

Continuous variables will be expressed as mean ± standard deviation, and categorical variables as frequencies and percentages.

Statistical analyses will include:

Wilcoxon signed-rank test: for within-group comparisons (baseline vs. 90-day values).

Mann-Whitney U test: for between-group comparisons.

Correlation analyses: between periodontal parameters (PPD, CAL, BOP) and renal markers (SCr, BUN, eGFR).

Significance level: p ≤ 0.05. Both per-protocol (PPA) and intention-to-treat (ITT) analyses will be performed to ensure robustness of findings.

Ethical Considerations

The study protocol has been reviewed and approved by the Institutional Review Board (IRB) of Dow University of Health Sciences. Written informed consent will be obtained from all participants prior to enrollment, with separate consent forms in English and Urdu to ensure understanding.

Participation is voluntary, and subjects may withdraw at any stage without penalty. All laboratory and dental procedures will be conducted free of cost. Participants in the control group will receive their complete periodontal therapy after the trial. Data confidentiality will be maintained through de-identification and restricted access.

Potential risks include mild discomfort during blood sampling and transient tooth sensitivity following SRP, both of which are minor and self-limiting. No major adverse effects are anticipated. Participants will have access to dental and medical support throughout the study period.

Expected Outcomes

The study anticipates a measurable improvement in renal function biomarkers (reduction in SCr and BUN levels, and improvement in eGFR) among the NSPT group compared to controls after 90 days. This would support the hypothesis that periodontal inflammation contributes to systemic inflammatory load affecting renal physiology.

Findings will help strengthen the understanding of oral-systemic health connections and may encourage multidisciplinary management of diabetic patients involving both dental and medical professionals.

Scientific Significance and Future Implications

This trial will be one of the first interventional studies from Pakistan evaluating the impact of non-surgical periodontal therapy on renal function in uncontrolled diabetics. The results could:

Provide evidence to include periodontal screening as part of diabetes management protocols.

Support collaborative programs between diabetology and dental departments for early detection and management of oral infections.

Encourage larger multicentric clinical trials exploring the long-term effects of periodontal therapy on renal and systemic outcomes in diabetic populations.

The study's integration of oral health and systemic disease management aligns with global efforts to promote interdisciplinary healthcare and may contribute to policy-level recommendations for diabetic patient care.

ELIGIBILITY:
Inclusion Criteria:

Adults between 30 and 65 years of age.

Men and women previously diagnosed with type 2 diabetes mellitus for at least one year.

Participants with uncontrolled diabetes, defined as HbA1c ≥ 7%.

Presence of moderate to severe gum disease (Stage II or Stage III periodontitis) as determined by a dental examination.

Estimated glomerular filtration rate (eGFR) of 60 mL/min/1.73 m² or higher.

Willing and able to provide written informed consent.

Exclusion Criteria:

Critically ill individuals or those unable to communicate effectively.

Pregnant or breastfeeding women.

Women currently using hormone replacement therapy or oral contraceptives within the past six months.

Individuals taking steroidal, nonsteroidal anti-inflammatory drugs (NSAIDs), or other anti-inflammatory medications within the past three months (except low-dose aspirin up to 75 mg daily).

Participants with a recent history of major blood loss, trauma, or gastrointestinal bleeding.

Use of antibiotics within the last month.

History of fever or vomiting lasting more than one week within the last month.

Regular tobacco or alcohol users.

Individuals with any other chronic disease or condition that could interfere with study outcomes.

Individuals unwilling or unable to comply with study procedures or follow-up visits.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Serum Creatinine, Blood Urea Nitrogen, and Estimated Glomerular Filtration Rate (eGFR) at 90 Days After Non-Surgical Periodontal Therapy | Baseline and 90 days after completion of non-surgical periodontal therapy
  The primary outcome will be evaluated by measuring changes in renal function biomarkers, including serum creatinine (mg/dL), blood urea nitrogen (BUN, mg/dL), and estimated glomerular filtration rate (eGFR, mL/min/1.73 m²). These parameters will be assessed at baseline and 90 days post-intervention to determine within- and between-group differences. Serum creatinine and BUN will be analyzed using standard automated laboratory methods, and eGFR will be calculated using the Modification of Diet in Renal Disease (MDRD) equation. A reduction in serum creatinine and BUN levels and an increase in eGFR will indicate improvement in renal function. Data will be statistically analyzed using Wilcoxon signed-rank and Mann-Whitney U tests with a significance threshold of p ≤ 0.05

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Scinces, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided